CLINICAL TRIAL: NCT05233449
Title: Nociception Level Index (NoL) Variation After Standardized Stimulation Under General Anesthesia in Children
Brief Title: NoL Index Response to Stimulation in Anesthetized Children
Acronym: STIMNOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021_0434; 2021-A02797-34 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia
Keywords: General anesthesia; Nociception; Monitoring; Nociception level; NoL

STUDY DESIGN:
Intervention Model Description: In order to avoid the bias related to the order of the stimuli, the order of application of the stimuli will be randomized according to a Latin square of order 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children anesthetized (Experimental): Inhalatory general anesthesia with sevoflurane 0.9 Minimal Alveolar Concentration and alfentanil 10 µg/kg
  Interventions: Device: NoL monitor; Procedure: Stimulation

INTERVENTIONS:
Device: NoL monitor — NoL monitor : non invasive, adhesive digital device
Procedure: Stimulation — Stimulation : 100 Hertz, 5 seconds, 10-30-60 milliamps, inner forearm

SUMMARY:
The Nociception Level (NoL) is an index obtained via a non-invasive monitor, that is currently used to assess nociception in anesthetized adults. The NoL index varies from 0 to 100. It increases in response to nociceptive stimuli. The objective of this study was to investigate if the NoL index also indicates the level of nociception in anesthetized children. In children anesthetized according to standard practice, before surgical incision, three 5-seconds stimulations will be performed with different intensities (10, 30 and 60 milliamps). The order of the stimulations intensities will be randomized. The hypothesis of study is that the intensity of stimulation will influence the magnitude of NoL-index increase in response to the stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-12 years
* Elective surgery under general anesthesia
* Written informed consent

Exclusion Criteria:

* Cardiac surgery
* Opioid intake < 24 hours before surgery
* Cardiac arrhythmia
* Pace maker
* Pheochromocytoma
* Anti-arrhythmic medication
* Anticholinergic medication
* Raynaud syndrome
* Digital anomaly (malformative, traumatic)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
NoL variation = [(Maximal NoL value in the 5 minutes following the stimulation) - (NoL before stimulation)] / [NoL before stimulation] | 5 minutes after stimulation
  NoL variation = [(Maximal NoL value in the 5 minutes following the stimulation) - (NoL before stimulation)] / [NoL before stimulation]

SECONDARY OUTCOMES:
Systolic Blood Pressure (SBP) variation | 5 minutes after stimulation
  SBP variation = [(Maximal SBP value in the 5 minutes following the stimulation) - (SBP before stimulation)] / [SBP before stimulation]
Analgesia Nociception Index (ANI) variation | 5 minutes after stimulation
  ANI variation = [(ANI before stimulation - (Minimal ANI value in the 5 minutes following the stimulation)] / [ANI before stimulation]

CONTACTS AND LOCATIONS:
Overall Officials: Nada Sabourdin, MD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Hopital Roger Salengro, CHU Lille, Lille
  - Hu Est Parisien Site Trousseau Aphp, Paris

REFERENCES:
- [Result] Chemam S, Cailliau E, Bert D, Tavernier B, Constant I, Sabourdin N. Nociception level response to calibrated stimulations in children: First assessment of the nociception level index in pediatric anesthesia. Anaesth Crit Care Pain Med. 2023 Jun;42(3):101207. doi: 10.1016/j.accpm.2023.101207. Epub 2023 Mar 1. PMID 36863410